CLINICAL TRIAL: NCT01652625
Title: Efficacy and Safety Study of Yunnan Baiyao on Minor Recurrent Aphthous Stomatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaosong Liu, associate professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peking University
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Yunnan Baiyao; recurrent aphthous stomatitis; clinical trial
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yunnan Baiyao toothpaste (Experimental): The toothpaste containing 6.5 milligrams of Yunnan Baiyao was used twice daily as part of the patient's routine oral hygiene for 5 days.
  Interventions: Drug: Yunnan Baiyao toothpaste
- placebo toothpaste (Active Comparator): One gram of placebo toothpaste was used twice daily by the control group patients. Except for the active Yunnan Baiyao extract, all ingredients contained in the placebo-toothpaste were the same as that in the experimental toothpaste.
  Interventions: Drug: Placebo toothpaste

INTERVENTIONS:
Drug: Yunnan Baiyao toothpaste — The patients were instructed to brush the teeth twice daily for 5 days, using 1 gram of Yunnan Baiyao toothpaste (equivocal to approximately 6-7 lines on a standard toothbrush) for 3 minutes. 6.5 milligrams of Yunnan Baiyao active extract were contained in 1 gram of the toothpaste.
  Arms: Yunnan Baiyao toothpaste
Drug: Placebo toothpaste — One gram of the placebo toothpaste was used twice daily by the control group patients. Except for the active Yunnan Baiyao extract, all ingredients contained in the placebo-toothpaste were the same as that in the experimental toothpaste.
  Arms: placebo toothpaste

SUMMARY:
Recurrent aphthous stomatitis (RAS) is a common recurrent oral disorder with no curative treatment available to date. The challenge remains in patients that do develop drug resistance and/or secondary infection, although topical corticosteroids and antimicrobials are the first therapeutic choice. The aim of the study was to evaluate the efficacy and safety of an herbal extract of Yunnan Baiyao formulated in toothpaste as an alternative therapy for minor RAS.

Yunnan Baiyao is a well-known traditional Chinese medicine, formulated in a powder or capsule form. It was initially and widely used in wounds for its anti-hemorrhagic hemostatic function, and further in gastrointestinal bleeding. Yunnan Baiyao powder has been generally applied on RAS among Chinese population.

In this study, a randomized, double-blind, placebo-controlled clinical trial (from March 2010 to March 2011) was conducted on a cohort of 227 minor RAS patients. The toothpaste containing Yunnan Baiyao was used twice daily as part of the patient's routine oral hygiene for 5 days. An assessment of ulcerative size and pain was recorded on Day 0 (baseline), Day 3 and Day 5. Any noted adverse reactions were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female aged 18 to 65 years old;
2. Patients diagnosed as minor recurrent aphthous stomatitis with the duration of each ulcer in excess of 5 days;
3. Fresh ulcers available with less than 72 hours eruption.

Exclusion Criteria:

1. Hypersensitive to various medical agents;
2. Concurrent acute infectious disease;
3. Pregnancy or lactation;
4. Concurrent other immunology disorders;
5. Accepting systemic administration of corticosteroids or immunosuppressive agents within 3 months;
6. Aphthous-like ulcers related to certain systemic disorders such as ulcerative colitis, Crohn's disease, Behcet's syndrome, serious anemia;
7. Aphthous-like ulcers related to drug such as non-steroidal anti-inflammatory drugs (NSAIDs) and anti-histamines;
8. Accepting anaesthetic therapy within 24 hours, or systemic antibiotics within 2 weeks, or other management for oral ulcers within 72 hours prior to the study;
9. Neoplasm patients;
10. Volunteers of other clinical trials on medical agents or toothpaste within one month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Ulcer size | one year
  The assessment of the surface area of the ulcer was measured in millimeters by a dental probe. Ulcer size was assessed as the product of maximum diameter and its vertical diameter.

SECONDARY OUTCOMES:
Pain Scores with Visual Analog Scale | one year
  Pain intensity was measured using a VAS, where the amount of pain recorded ranged from 0 (no pain) to 10 (unbearable pain). Pain was assessed by irritating the ulcer with the periodontal probe. The values were collected by the assigned investigators.
Number of the participants with adverse events | one year
  Any noted adverse reactions were recorded.